CLINICAL TRIAL: NCT03014817
Title: Ultrasonically Activated Scalpel Versus Electrocautery Based Dissection in Acute Cholecystitis. A Randomized, Double Blind, Multicenter Study
Brief Title: Ultrasonically Activated Scalpel Versus Electrocautery Based Dissection in Acute Cholecystitis Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Gabriel Sandblom, Associate Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Ultrasonic scalpel trial
Record Dates: First submitted 2017-01-05; First posted 2017-01-09 (Estimated); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Cholecystitis, Acute
MeSH Terms: conditions — Cholecystitis, Acute | interventions — Electrocoagulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasonically activated scalpel (Experimental): Dissection with ultrasonically activated scalpel. Direction of dissection undecided but by experience most naturally fundus first.
  Interventions: Procedure: Ultrasonically activated scalpel
- Electrocautery (Active Comparator): Dissection with electrocautery. Direction of dissection undecided but by experience most naturally cystic duct first.
  Interventions: Procedure: Electrocautery

INTERVENTIONS:
Procedure: Ultrasonically activated scalpel — Dissection with ultrasonically activated scalpel
  Arms: Ultrasonically activated scalpel
Procedure: Electrocautery — Dissection with electrocautery
  Arms: Electrocautery

SUMMARY:
The present study aims at analyzing whether ultrasonic tissue coagulation dissection technique offers a smoother peri- and postoperative course and reduces the risk for conversion from laparoscopic to open surgery in acute cholecystectomy patients as compared to electrocautery in case of acute cholecystitis The study is performed as a double-blinded study on patients undergoing laparoscopic surgery for acute cholecystitis. Patients included in the study are randomized to surgery with either the traditional electrocautery based technique or ultrasonic scalpel based dissection.

DETAILED DESCRIPTION:
Electrocautery is traditionally the method of choice for tissue dissection in laparoscopic cholecystectomy. As an alternative to electrocautery, the ultrasonically activated scalpel has proven to be an effective and safe instrument for the facilitation of dissection and to minimize blood loss in both open and laparoscopic surgery. Whereas electrocautery coagulates by burning at temperatures higher than 150ºC, the ultrasonic scalpel transforms the electric power into mechanical longitudinal vibration of the working part of the instrument by a piezoelectrical transducer. Accordingly, the former technique limits the heating- thermal necrosis effect on the tissue to the area just adjacent to the cutting line.

Since the relative-potential benefit of the ultrasonic scalpel is high in technically demanding surgery, the advantage may not be as pronounced in routine laparoscopic gallstone surgery, which can usually be done more uneventfully whichever equipment is used. Laparoscopic cholecystectomy for acute cholecystitis is, however, more demanding connected with longer operative time, more postoperative complications, greater risk of conversion to open cholecystectomy and longer postoperative stay. In addition, we know that operations for acute cholecystitis are associated with a higher risk for severe complications such as bile duct injury. The potential benefit from using the ultrasonic scalpel is thus even greater when doing surgery for cholecystitis.

In addition to this there are numerous important aspects on the safety in the implementation of the emergency cholecystectomy. Traditionally, most surgeons have chosen to operate these patients with laparoscopic technique, with the use of a so-called electrocautery hook, which usually allows tissue division with minimal blood loss. Further improvements in the dissection technique followed the introduction of ultrasonic tissue coagulation. This technique offers the option of performing these operations with even less blood loss, a more gentle handling of the inflamed tissue and a sealing of the tissue sections while the tissue is divided. Accordingly this ultrasonic tissue coagulation technique can theoretically be of significant advantage not the least when dividing acutely inflamed tissue like in acute cholecystitis with particular relevance for the dissection of the gallbladder from the liver bed, where bleeding and bile leakage often occurs. Moreover if the surgeon instead chooses to dissect the gallbladder from the doom and downwards, to the part that contains the cystic duct and cystic artery (Calots triangle), unique options can be offered to not only simplify the operation but also make it safer. This latter technique is called "fundus first".

The present study aims at analyzing whether ultrasonic tissue coagulation dissection technique combined with "fundus first" approach offers a smoother per and postoperative course in acute cholecystectomy patients as compared to the traditional way of performing the operation. Due to the lower risk of bleeding and better anatomical overview, the technique may also reduce the risk of having to convert the procedure for laparoscopic cholecystectomy to open cholecystectomy.

The study is performed as a double-blinded study on patients undergoing laparoscopic surgery for acute cholecystitis. Patients included in the study are randomized to surgery with either the traditional electrocautery based technique or ultrasonic scalpel based dissection with the "fundus first" approach.

The choice of dissection approach is determined by the randomization procedure, whether it is done from the triangle of Callot + electrocautery and upwards or from the gallbladder fundus and downwards by the use of the ultrasonic scalpel. Peroperative cholangiography is done routinely. The cystic duct is closed with a clip, not with the ultrasonic scalpel.

One month after surgery the patient is contacted by a telephone. In cases the questionnaires have not been returned yet, the patient is reminded about this. At the phone call the exact number of days of sick leave postoperatively and any adverse events occurring after discharge are recorded.

ELIGIBILITY:
Inclusion Criteria:

* Emergency laparoscopic cholecystectomy performed for cholecystitis
* American Society of Anesthesiologists (ASA) score I-III

Exclusion Criteria:

* Patients unable to express themselves in Swedish
* Pregnancy
* Previous open surgery in the upper abdomen
* American Society of Anesthesiologists (ASA) score >III

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2023-03-22 (Actual); Study Completion 2023-03-22 (Actual)

PRIMARY OUTCOMES:
Postoperative complications | 30 days
  Postoperative complications registered according to Clavien-Dindo

SECONDARY OUTCOMES:
Operative time | 3 hours
  Time required to complete surgery
Level of technical complexity | 3 hours
  Level of technical complexity of the procedure as assessed by the surgeon
Technical performance | 3 hours
  Perioperative technical performance assessed by an independent observer
Postoperative stay | 14 days
  Time from surgery to duscharge
Sick leave | 30 days
  Time from surgery to return to work
Conversion rate | 3 hours
  Conversion from laparoscopic to open cholecystyectomy
Postoperative pain | 7 days
  Daily assessments of pain on a visual analogue scale
Postoperative inflammatory activity | 7 days
  Daily measurements of c-reactive protein and leukocyte particle concentration
Conversion rate | 3 hours
  Number of procedures converted to open cholecystectomy
Direct and indirect medical costs | 30 days
  Analysis of health economics

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Sandblom, Assoc Prof, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska University Hospital, Center for Digestive Diseases, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Blohm M, Sandblom G, Enochsson L, Cengiz Y, Bayadsi H, Hennings J, Diaz Pannes A, Stenberg E, Bewo K, Osterberg J. Ultrasonic dissection versus electrocautery dissection in laparoscopic cholecystectomy for acute cholecystitis: a randomized controlled trial (SONOCHOL-trial). World J Emerg Surg. 2024 Nov 13;19(1):34. doi: 10.1186/s13017-024-00565-4. PMID 39538278